CLINICAL TRIAL: NCT02888093
Title: A Randomized Controlled Trial of Permanent vs Absorbable Suture for Uterosacral Ligament Suspension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Kowalski (Other)
Collaborators: International Urogynecological Association (Other)
Responsible Party: Sponsor-Investigator, Joseph Kowalski, Female Pelvic Medicine and Reconstructive Surgery, Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201607769
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Pelvic Organ Prolapse; Cystocele; Uterine Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absorbable (Experimental): Absorbable suture (polydioxanone) for uterosacral ligament suspension (USLS)
  Interventions: Device: Absorbent suture (polydioxanone) and Permanent suture (Gore-Tex CV2)
- Permanent (Experimental): Permanent suture (Gore-Tex CV2) for uterosacral ligament suspension (USLS)
  Interventions: Device: Absorbent suture (polydioxanone) and Permanent suture (Gore-Tex CV2)

INTERVENTIONS:
Device: Absorbent suture (polydioxanone) and Permanent suture (Gore-Tex CV2)

SUMMARY:
Uterosacral ligament suspension (USLS) is a commonly performed, vaginal surgery for the correction of female pelvic organ prolapse. The original description of this procedure included the use of permanent sutures. However, permanent suture use in this vaginal application can result in some minor complication such as persistent vaginal spotting, vaginal discharge and dyspareunia. Subsequent reports on this procedure have utilized delayed-absorbable sutures in order to avoid these complications. Retrospective studies are conflicting as to whether or not absorbable suture provides as durable an anatomic outcome as permanent suture. There are currently no high-quality, prospective studies that have evaluated outcomes of permanent and absorbable suture for uterosacral ligament suspension.

This study will recruit women scheduled to undergo USLS with or without other prolapse or anti-incontinence procedures. Participants will be randomized 1:1 to permanent or absorbable suture. Follow up will occur at 6 weeks and 12 months post-operatively. The primary outcome will be Pelvic Organ Prolapse Quantification Exam (POP-Q) point C as measured at the 12 month follow up visit. Subjects and assessors will be blinded.

DETAILED DESCRIPTION:
Patient demographics, relevant histories, baseline physical exam including POP-Q and PFDI-20 data will be abstracted from the electronic medical record following enrollment. This information will be placed into a secure database.

The randomization sequence will be generated by randomize.net, a web-based service that provides comprehensive randomization services for randomized controlled trials. The sequence will be randomized 1:1 with blocks of 4 and stratified by surgeon. Concealment will be completely opaque as group allocation will not be revealed until the subject is enrolled on the web-based service and the surgeon has elected to randomize the patient from an internet connection in the operating room.

Subjects and assessors will be blinded to study group. The surgeons will, necessarily, not be blinded. Subjects will only be informed of their assigned group upon request following completion of the entire study.

USLS with the assigned suture and any scheduled concomitant prolapse and anti-incontinence procedures will be performed. All procedures will be performed by one of two fellowship-trained, Female Pelvic Medicine and Reconstructive Surgery board-certified surgeons. USLS will be performed as initially described by Shull et al with two important differences in technique. First, 2 sutures will be placed through the intermediate portion of each uterosacral ligament instead of 3. Second, when absorbable suture (polydioxanone) is used, the suture will be placed through the full thickness of the anterior and posterior vaginal walls.

Follow up exams will occur at 6 weeks and 12 months post-operatively and will include a POP-Q exam. The 6 week follow up visit will include the Patient Global Impression of Improvement (PGI-I) and an additional survey. The 12 month follow up visit will include a the PGI-I, PFDI-20 and an additional survey. All participants will also be assessed for any suture-related complications, such as erosion or granulation tissue. Follow up exams will be completed by one of two urogynecology nurse practitioners who will be blinded to the surgery and suture choice. Both nurse practitioners have extensive experience in performing POP-Q exams. The examiners will complete a follow up data abstraction form for each follow up appointment (6 weeks and 12 months).

The follow up clinic appointments at 6 weeks and 12 months are the times of usually scheduled post-operative follow up for USLS procedures. Additionally, completion of the PFDI-20 questionnaire and a POP-Q exam constitute routine clinical care for these patients. As such, there is no additional time commitment for subjects compared to routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for uterosacral ligament suspension (USLS)

Exclusion Criteria:

* Non-English speaking
* Prisoner
* Cognitive impairment precluding informed consent
* Planned hysteropexy

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Kowalski, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Absorbable: Absorbable suture (polydioxanone) for uterosacral ligament suspension (USLS)
  Absorbent suture (polydioxanone) and Permanent suture (Gore-Tex CV2)
- Permanent: Permanent suture (Gore-Tex CV2) for uterosacral ligament suspension (USLS)
  Absorbent suture (polydioxanone) and Permanent suture (Gore-Tex CV2)
Period: Overall Study
Arm/Group | Absorbable | Permanent
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorbable | Permanent | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (13.7) | 63.6 (10.2) | 62.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Pelvic Organ Prolapse Quantification Exam (POP-Q) Point C
Description: Non-inferiority of POP-Q point C. This measure was obtained as originally described by Bump et al. The hymen is used as a fixed reference point. In other words, this is point zero. Point C is measured in cm relative to the hymen with negative values being proximal to the hymen and positive values distal to the hymen. Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy.
Time Frame: 12 months
Measure: Median (Full Range); unit: cm
Arm/Group | Absorbable | Permanent
Number analyzed (Participants) | 20 | 20
cm | -7.25 [-9 to -5.5] | -7 [-10 to -6]

2. Secondary Outcome: Suture-related Complications
Description: The presence of apical granulation tissue, apical suture exposure, abnormal vaginal discharge, vaginal spotting, post-coital spotting, dyspareunia or patient being able to feel suture.
Time Frame: 6 weeks and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Absorbable | Permanent
Number analyzed (Participants) | 20 | 20
Participants
  6 weeks | 17 | 14
  12 months | 2 | 4

3. Secondary Outcome: Symptomatic Prolapse Outcomes
Description: Positive response to PFDI-20 question #3 regarding the presence of a vaginal bulge (yes) AND the presence of bother (somewhat, moderately or quite a bit).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Absorbable | Permanent
Number analyzed (Participants) | 20 | 20
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Absorbable | Permanent
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 2/22 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absorbable (N=22) | Permanent (N=22)
Any suture related complication (Reproductive system and breast disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT02888093/Prot_000.pdf